CLINICAL TRIAL: NCT04148209
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED STUDY TO ASSESS THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE ASCENDING ORAL DOSES OF PF-07081532 IN HEALTHY ADULT PARTICIPANTS
Brief Title: Study of Single Ascending Doses of PF-07081532 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C3991001; 2019-003012-30 (EudraCT Number)
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: First-in-human study

STUDY DESIGN:
Intervention Model Description: This study is a double-blinded (investigator- and participant-blinded), sponsor-open, randomized, single-ascending oral dose, 4-period crossover, placebo substitution design in 2 interleaving cohorts of healthy adult participants. An additional cohort, enrolling healthy adult participants in up to 4 crossover periods, may be included to permit assessment of any of the following: repeat of a previously administered dose level; studying additional dose levels as dictated by the evaluated safety, tolerability or PK of earlier dose levels; or any other assessment needed to meet the objectives of this study. A cohort enrolling Japanese participants to receive PF-07081532 or placebo in up to 3 periods, may be included.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants receiving PF-07081532
  Interventions: Drug: PF-07081532
- Placebo (Placebo Comparator): Participants receiving Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07081532 — Participants will receive single ascending doses PF-07081532
  Arms: Treatment
Drug: Placebo — Participants will receive placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of single ascending oral doses of PF-07081532 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female (of non-childbearing potential) participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, including blood pressure (BP) and pulse rate measurement, temperature, standard 12-lead ECG, telemetry and laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures. Note that participants enrolling as Japanese must have 4 biological Japanese grandparents who were born in Japan.
4. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in the protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal (including pancreatitis), cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
3. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing at screening for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis B surface antibody (HBsAb) or hepatitis C antibody (HCVAb).
4. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2), or participants with suspected MTC per the investigator's judgement.
5. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
6. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
7. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).
8. A positive urine drug test at screening or admission.
9. Screening supine BP >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest.
10. Screening standard 12-lead single ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline Fridericia-corrected QT [QTcF] interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias).
11. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >=1.25 × upper limit of normal (ULN); total bilirubin level >=1.5 × ULN, participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <= ULN; TSH > ULN; HbA1c >= 6.5%.
12. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
13. Use of tobacco/nicotine containing products more than 5 cigarettes/day.
14. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
15. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of the protocol.
16. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events | From screening until follow-up call (28-35 days after the last dose of investigational product)
Percentage of participants with safety laboratory test results above/below certain threshold | Days -1, 2 and 4 of each period and at follow-up visit (7-14 days after the last dose of investigational product)
Percentage of participants with vital signs above/below certain threshold | Days 1-4 of each period and at follow-up visit (7-14 days after the last dose of investigational product)
Percentage of participants with 12-lead electrocardiogram (ECG) results above/below certain threshold | Days 1-4 of each period and at follow-up visit (7-14 days after the last dose of investigational product)

SECONDARY OUTCOMES:
PF-07081532 AUClast | Days 1-4 of each period
  Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration
PF-07081532 AUCinf | Days 1-4 of each period
  Area under the plasma concentration-time profile from time 0 extrapolated to infinite time
PF-07081532 Cmax | Days 1-4 of each period
  Maximum plasma concentration
PF-07081532 Tmax | Days 1-4 of each period
  Time for maximum plasma concentration
PF-07081532 t1/2 | Days 1-4 of each period
  Terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991001